CLINICAL TRIAL: NCT05609175
Title: Investigating the Relationship Between Nocturnal Glucose Levels and Motion During Sleep - The Moonwalk Pilot-Study
Brief Title: Investigating the Relationship Between Nocturnal Glucose Levels and Motion During Sleep
Acronym: Moonwalk
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); DCB Research AG (Other)
Responsible Party: Sponsor
Other Study IDs: Moonwalk Pilot
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Diabetes; Hypoglycemia; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study the investigators will explore whether the motion during sleep of people with diabetes changes as a function of the blood glucose levels. The motion will be assessed with a radar sensor, a thermal camera, and wrist worn smartwatches. Additionally, participants will answer a short daily questionnaire. Data will be collected for 10 days and analyzed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Age ≥ 18 years
* Patients at the outpatient clinics or from a referring diabetologist with a diagnostic CGM according to best medical practice
* Patients with diabetes mellitus on an insulin therapy or with non-insulin antidiabetic medication with the potential to induce hypoglycemia
* HbA1c value between 6% and 10% (inclusive) within 6 months prior to inclusion

Exclusion Criteria:

* Wearables cannot be attached around the wrist of the patient
* Known allergies to components of the wearables
* Female subjects: pregnancy, lactation period, lack of a negative urine pregnancy test (except in case of menopause, sterilization or hysterectomy), or unwilling to use a contraception during the study (for sexually active subjects of childbearing potential)
* Known cardiac arrhythmia (e.g., atrial flutter or fibrillation, Atrioventricular-reentry tachycardia, Atrioventricular block > grade 1)
* Pacemaker or ICD (implantable cardioverter defibrillator)
* Treatment with antiarrhythmic drugs or beta-blockers
* Drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
* Any illness or use of medications that could affect sleep patterns (including sleep apnea)
* Dependency from the sponsor or the clinical investigator
* Participation in another investigation with an investigational drug or a pre-market medical device within the 30 days preceding and during the present investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 or type 2 diabetes mellitus on an insulin therapy or with non-insulin antidiabetic medication.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Area under the receiver operator characteristics curve (AUROC) in detecting nocturnal level 1 hypoglycemia based on motion data obtained by radar signals | For the entire wear time of the diagnostic continuous glucose monitor (CGM), up to 10 days
  Level 1: glucose < 3.9 mmol/L
  Motion data obtained from radar signals

SECONDARY OUTCOMES:
Correlation coefficient between nocturnal glucose levels and motion | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Nocturnal glucose will be measured with a CGM and motion will be measured with the radar signal as average dispersion index across all range bins in the range-doppler map
Correlation coefficient between nocturnal glucose levels and motion | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Nocturnal glucose will be measured with a CGM and motion will be measured with the radar signal as the average of detected points in the 3D point cloud from the radar sensor
Correlation coefficient between nocturnal glucose levels and physiological data | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Nocturnal glucose will be measured with a CGM and physiological data, i.e., heart rate, heart rate variability, respiratory rate, will be gathered from smartwatches.
Correlation coefficient between nocturnal glucose levels and physiological data and radar data | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Nocturnal glucose will be measured with a CGM and physiological data, i.e., heart rate, heart rate variability, respiratory rate, will be gathered from smartwatches. Motion will be measured with the radar signal as the average dispersion index across all range bins in the range-doppler map or the average of detected points in the 3D point cloud from the radar sensor
Time spent in euglycemia | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Glucose will be measured with a CGM. Euglycemia is defined as 4.0 - 10.0 mmol/L. The time will be illustrated as percent of CGM measurements within this range.
Time spent below 3.9 mmol/L | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Glucose will be measured with a CGM. The time will be illustrated as percent of CGM measurements.
Time spent below 3.0 mmol/L | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Glucose will be measured with a CGM. The time will be illustrated as percent of CGM measurements.
Time spent above 10.0 mmol/L | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Glucose will be measured with a CGM. The time will be illustrated as percent of CGM measurements.
Time spent above 13.9 mmol/L | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Glucose will be measured with a CGM. The time will be illustrated as percent of CGM measurements.
Course of nocturnal glucose levels | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Glucose will be measured with a CGM in mmol/L
Course of nocturnal motion according to thermal camera measurements | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Glucose will be measured with a CGM and thermal camera measurements
Course of nocturnal hypoglycemia symptoms according to thermal camera measurements and/or physiological data | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
Glucose level at start of hyperglycemia symptoms | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Measured by CGM
Glucose level at start of hypoglycemia symptoms | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Measured by CGM
AUROC in detecting nocturnal hyperglycemia based on motion data (radar signals) | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Glucose > 10.0 mmol/L
AUROC in detecting nocturnal level 2 hypoglycemia based on motion data | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Glucose < 3 mmol/L
  Motion data extracted from radar signals
AUROC in detecting nocturnal hyperglycemia, nocturnal level 1 and level 2 hypoglycemia based on motion data, physiological data, and Artificial Intelligence | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Level 1: glucose < 3.9 mmol/L
  Level 2: glucose < 3 mmol/L motion data extracted from radar signals
AUROC in classifying nocturnal dysglycemia symptoms based on motion data, physiological data, and Artificial Intelligence | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Dysglycemia: <4.0 and >10.0 mmol/L
  Motion data extracted from radar signals
AUROC in classifying motion patterns according to thermal camera measurements based on motion data, physiological data, and Artificial Intelligence | For the entire wear time of the diagnostic continuous glucose monitor, up to 10 days
  Motion data extracted from radar signals

CONTACTS AND LOCATIONS:
Overall Officials: Markus Laimer, Prof.Dr.med., Principal Investigator — Inselspital; Lilian Witthauer, Prof.Dr., Study Director — University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Inselspital Bern, University and University Hospital Bern, Bern, Switzerland